CLINICAL TRIAL: NCT01756807
Title: Evaluation of Endothelial ProGenitor Cell Capture Sirolimus-Eluting Stent by Optical Coherence Tomography: the COMBO Stent Angiographic Extension Study (EGO-COMBO Angiographic Extension Study)
Brief Title: EGO-COMBO Angiographic Extension Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Stephen Lee (Other)
Responsible Party: Sponsor-Investigator, Prof. Stephen Lee, Professor and Chief, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 12-472 (IRB HK)
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Coronary Disease
Keywords: Optical Coherence Tomography; Geneous Stent; Combo Stent
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- The Combo Stent (Experimental): The COMBO Stent is developed basing on the GENOUS stent platform, and in addition, it also delivers a drug called sirolimus to the treated coronary blood vessel. The stent's original CD34 antibody coating is designed to promote healing of the coronary artery by catching circulating endothelial progenitor cells as they pass through the stent. These cells are naturally flowing in the circulation and are responsible for endothelial healing. This is intended to help the blood vessel wall heal over the stent more quickly and restore normal tissue function in the stented area. The combination of these two technologies in this new COMBO stent is expected to produce even better clinical results, which have been investigated in the previous REMEDEE Study.
  Interventions: Device: The COMBO Stent

INTERVENTIONS:
Device: The COMBO Stent — The COMBO Stent is developed basing on the GENOUS stent platform, and in addition, it also delivers a drug called sirolimus to the treated coronary blood vessel. The stent's original CD34 antibody coating is designed to promote healing of the coronary artery by catching circulating endothelial progenitor cells as they pass through the stent. These cells are naturally flowing in the circulation and are responsible for endothelial healing. This is intended to help the blood vessel wall heal over the stent more quickly and restore normal tissue function in the stented area. The combination of these two technologies in this new COMBO stent is expected to produce even better clinical results, which have been investigated in the previous REMEDEE Study.

SUMMARY:
Evaluation of Endothelial ProGenitor Cell Capture Sirolimus-Eluting Stent by Optical Coherence Tomography: the COMBO Stent angiographic extension Study (EGO-COMBO angiographic extension Study)

DETAILED DESCRIPTION:
The Genous Stent (the EPC Capture R-stent, OrbusNeich Medical Inc., Fort Lauderdale, FL) is commercially available and has been used extensively in standard coronary intervention in the treatment of more than 200 patients with critical coronary stenoses at Queen Mary Hospital. The COMBO Stent (OrbusNeich Medical Inc., Fort Lauderdale, FL) is an improved version of the Genous Stent and has been implanted in 60 patients at Queen Mary Hospital. All patients have remained in good condition since the treatment.

The Genous Stent is a bio-engineered 316L stainless steel coronary stent with a biocompatible coating having specific CD34 antibody on the inner surface. CD34 is a surface antigen present on circulating endothelial progenitor cell (EPC). It will be bonded to the CD34 antibody, resulting in capturing of the EPC onto the stent surface and differentiation into endothelial layer. Animal model has demonstrated that a functional endothelial layer could be formed as soon as 24 to 48 hours after Genous stent implantation (1). The HEALING-FIM registry has shown that Genous stent is clinically safe and effective in the treatment of coronary stenosis (2). Recent reports have further confirmed its efficacy in patients with acute coronary syndrome requiring urgent revascularization (3,4).

The COMBO Stent is developed basing on the GENOUS stent platform, and in addition, it also delivers a drug called sirolimus to the treated coronary blood vessel. The stent's original CD34 antibody coating is designed to promote healing of the coronary artery by catching circulating endothelial progenitor cells as they pass through the stent. These cells are naturally flowing in the circulation and are responsible for endothelial healing. This is intended to help the blood vessel wall heal over the stent more quickly and restore normal tissue function in the stented area. The combination of these two technologies in this new COMBO stent is expected to produce even better clinical results, which have been investigated in the previous REMEDEE Study.

Animal study has shown the COMBO Stent promotes endothelialization and reduces neointima formation, as assessed by both optical coherence tomography (OCT) and histopathology (5). Even though COMBO Stents have been used and found to be safe in over 210 patients world-wide and in about 61 patients at Queen Mary Hospital under the EGO-COMBO Study Protocol, such beneficial endothelial coverage as assessed by OCT has never been documented in human subjects.

This current EGO-COMBO angiographic extension study protocol is designed based on the approved protocol EGO-COMBO Study (IRB: UW 10-342). This current study mainly focuses on the time frame, degree of endothelialization, and the subsequent neointimal proliferation after COMBO Stent implantation from 2 years, as assessed by intracoronary optical coherence tomography (OCT).

Intracoronary optical coherence tomography (OCT) is a simple catheter-based imaging technique using optic fibre to achieve very detailed assessment (resolution down to 100 microns) in intra-coronary stent apposition, early stent coverage (endothelialization) and late stent neoinitmal growth (restenosis). It is performed as part of routine cardiac catheterization procedure and provides high-resolution cross sectional images of the coronary arteries. OCT has been shown to be safe in clinical practice (6, 7). The C7XR OCT system (Frequency Domain OCT) is a commercial available product with CE Mark and FDA approval. The OCT catheter is just a non-occlusive optic fibre which is extremely small and flexible and will pose no additional risk to the patient other than those inherent risks of a standard angioplasty procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-85 years old
* Patient who agrees to have follow-up coronary angiograms
* Patient who were previously enrolled in EGO-COMBO study

Exclusion Criteria:

* Patient who refuses to consent to coronary angiogram or coronary angioplasty

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Co-primary end-points of OCT findings on coverage (degree of endothelialization) and OCT findings on late loss (late tissue growth, plaque volume, lumen cross sectional area), binary restenosis and late angiographic late loss by QCA at two years restudy. | At the two year restudy date
  Co-primary end-points of OCT findings on coverage (degree of endothelialization) and OCT findings on late loss (late tissue growth, plaque volume, lumen cross sectional area), binary restenosis and late angiographic late loss by QCA at two years restudy.

SECONDARY OUTCOMES:
Any major adverse cardiac events at two years restudy. | At the two year restudy date.
  Any major adverse cardiac events at two years restudy.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen WL Lee, MD FRCP FACC, Principal Investigator — Department of Medicine, The University of Hong Kong, Queen Mary Hospital, Hospital Authority
Locations (1):
- Department of Medicine, the University of Hong Kong, Queen Mary Hospital, Hospital Authority, Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Alfonso F, Dutary J, Paulo M, Gonzalo N, Perez-Vizcayno MJ, Jimenez-Quevedo P, Escaned J, Banuelos C, Hernandez R, Macaya C. Combined use of optical coherence tomography and intravascular ultrasound imaging in patients undergoing coronary interventions for stent thrombosis. Heart. 2012 Aug;98(16):1213-20. doi: 10.1136/heartjnl-2012-302183. PMID 22826559
- [Background] Kutryk MJ, Kuliszewski MA. In vivo endothelial progenitor cell seeding for the accelerated endothelialization of endovascular devices. Am J Cardiol 2003; 92:94L
- [Background] Aoki J, Serruys PW, van Beusekom H, Ong AT, McFadden EP, Sianos G, van der Giessen WJ, Regar E, de Feyter PJ, Davis HR, Rowland S, Kutryk MJ. Endothelial progenitor cell capture by stents coated with antibody against CD34: the HEALING-FIM (Healthy Endothelial Accelerated Lining Inhibits Neointimal Growth-First In Man) Registry. J Am Coll Cardiol. 2005 May 17;45(10):1574-9. doi: 10.1016/j.jacc.2005.01.048. PMID 15893169
- [Background] Co M, Tay E, Lee CH, Poh KK, Low A, Lim J, Lim IH, Lim YT, Tan HC. Use of endothelial progenitor cell capture stent (Genous Bio-Engineered R Stent) during primary percutaneous coronary intervention in acute myocardial infarction: intermediate- to long-term clinical follow-up. Am Heart J. 2008 Jan;155(1):128-32. doi: 10.1016/j.ahj.2007.08.031. Epub 2007 Nov 26. PMID 18082503
- [Background] Miglionico M, Patti G, D'Ambrosio A, Di Sciascio G. Percutaneous coronary intervention utilizing a new endothelial progenitor cells antibody-coated stent: a prospective single-center registry in high-risk patients. Catheter Cardiovasc Interv. 2008 Apr 1;71(5):600-4. doi: 10.1002/ccd.21437. PMID 18360849
- [Background] Granada JF, Inami S, Aboodi MS, Tellez A, Milewski K, Wallace-Bradley D, Parker S, Rowland S, Nakazawa G, Vorpahl M, Kolodgie FD, Kaluza GL, Leon MB, Virmani R. Development of a novel prohealing stent designed to deliver sirolimus from a biodegradable abluminal matrix. Circ Cardiovasc Interv. 2010 Jun 1;3(3):257-66. doi: 10.1161/CIRCINTERVENTIONS.109.919936. Epub 2010 May 4. PMID 20442358
- [Background] Yamaguchi T, Terashima M, Akasaka T, Hayashi T, Mizuno K, Muramatsu T, Nakamura M, Nakamura S, Saito S, Takano M, Takayama T, Yoshikawa J, Suzuki T. Safety and feasibility of an intravascular optical coherence tomography image wire system in the clinical setting. Am J Cardiol. 2008 Mar 1;101(5):562-7. doi: 10.1016/j.amjcard.2007.09.116. Epub 2008 Jan 10. PMID 18307999
- [Background] Prati F, Cera M, Ramazzotti V, Imola F, Giudice R, Albertucci M. Safety and feasibility of a new non-occlusive technique for facilitated intracoronary optical coherence tomography (OCT) acquisition in various clinical and anatomical scenarios. EuroIntervention. 2007 Nov;3(3):365-70. doi: 10.4244/eijv3i3a66. PMID 19737719
- [Derived] Lee SW, Lam SC, Tam FC, Chan KK, Shea CP, Kong SL, Wong AY, Yung A, Zhang LW, Tse HF, Wu KK, Chan R, Haude M, Mehran R, Mintz GS, Maehara A. Evaluation of Early Healing Profile and Neointimal Transformation Over 24 Months Using Longitudinal Sequential Optical Coherence Tomography Assessments and 3-Year Clinical Results of the New Dual-Therapy Endothelial Progenitor Cell Capturing Sirolimus-Eluting Combo Stent: The EGO-Combo Study. Circ Cardiovasc Interv. 2016 Jul;9(7):e003469. doi: 10.1161/CIRCINTERVENTIONS.115.003469. PMID 27418609